CLINICAL TRIAL: NCT03475693
Title: A Cohort Study Evaluating the Efficacy of PO Magnesium in the Treatment of Acute Traumatic Brain Injury in Adolescents
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Corewell Health South (Other)
Collaborators: Michigan State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MMMC#1571
Record Dates: First submitted 2017-08-08; First posted 2018-03-23 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Concussion Post Syndrome
MeSH Terms: conditions — Post-Concussion Syndrome | interventions — Magnesium Oxide; Acetaminophen; Ondansetron

STUDY DESIGN:
Intervention Model Description: Randomized, prospective, cohort study comparing two non-invasive treatments for Mild traumatic brain injury in patients ages 12-18 that present to the Lakeland Health Emergency departments in either St. Joseph, MI or Niles, MI.
Who Masked: Participant
Masking Description: Patients will be assigned a 3 digit number given at random and treatment arm will be randomized to day of presentation with treatment determined by even or odd day of the month
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment arm (Experimental): Patients will receive PO magnesium 400 mg, Zofran 4 mgODT, and Tylenol 500 mg in the emergency department. They will then continue with 500 mg Tylenol BID and 400 mg MagOx tablets BID for the next 5 days. Symptom severity scores will be obtained and compared throughout this time as mentioned in the study design.
  Interventions: Drug: Magnesium Oxide; Drug: Acetaminophen; Drug: Zofran ODT 4 MG Disintegrating Oral Tablet
- Placebo arm (Placebo Comparator): Patients will receive PO Zofran 4 mgODT, and Tylenol 500 mg in the emergency department. They will then continue with 500 mg Tylenol BID for the next 5 days. Symptom severity scores will be obtained and compared throughout this time as mentioned in the study design.
  Interventions: Drug: Acetaminophen; Drug: Zofran ODT 4 MG Disintegrating Oral Tablet

INTERVENTIONS:
Drug: Magnesium Oxide — 400 mg Magnesium oxide tablet given once in the ED, and prescribed to take BID for 5 days total after discharge
  Arms: Treatment arm
Drug: Acetaminophen — 500 mg tablets given once in the ED, and prescribed to take BID for 5 days total after discharge.
Drug: Zofran ODT 4 MG Disintegrating Oral Tablet — Given once in the Emergency department

SUMMARY:
The objective of this study is to evaluate the efficacy of magnesium in symptomatic reduction of mild traumatic brain injury in the adolescent population in the acute setting of injury.

DETAILED DESCRIPTION:
Introduction Mild traumatic brain injuries are a growing problem in sports, and are now becoming publicly relevant. Mild traumatic brain injuries account for 700,000 ED visits, hospitalizations, and deaths annually. Today, 1 out of 5 adolescents will be affected by mild traumatic brain injuries. Magnesium is a critical neuromodulator that plays an important role in controlling neural signaling in the brain, and studies have shown a transiently low level of magnesium in CNS neurons following traumatic brain injury. If these electrolyte imbalances could be corrected with magnesium supplementation during the acute injury, this could potentially decrease the symptomatic period in those with mild TBI. The investigators aim to show a correlation between administration of PO magnesium and increased resolution of symptoms thereby improving the subjective recovery course of adolescents with concussion.

Study objective This randomized, cohort study will compare the clinical efficacy of PO magnesium and Zofran, to that of PO Tylenol and Zofran in the treatment of adolescents presenting within 48 hours of a mild traumatic brain injury.

Purpose With current studies and the sports media revolving around the long-term effects of repetitive mild TBI, it is important to continue to improve treatment of these injuries. Current therapy revolves around symptomatic care, rest, and return to school/sport after symptoms have resolved and the patient has been cleared by a physician. After a concussion, there is a period of 7-10 days where the patient has a transient decrease in the participants mental functioning. The investigators hope to decrease the length of the acute symptomatic period by supplementing oral magnesium along with the current symptomatic care. Studies have shown that IV magnesium in high doses can improve the function of patients with severe TBI. There have not been many studies looking at the efficacy of PO magnesium in this setting. While there is no evidence that concussions have long term effects on neurocognitive function, this study could add to the existing algorithm for concussion management.

Hypothesis The investigators believe that administration of magnesium in patients who present with mild traumatic brain injuries will decrease post concussive symptoms, thereby speeding recovery.

Methods Study design and setting Randomized, prospective, parallel cohort study comparing two non-invasive treatments for Mild traumatic brain injury in patients ages 12-18 that present to the Lakeland Health Emergency departments in either St. Joseph, MI or Niles, MI. The data collection period will take approximately 2 years with a minimum goal of 76 patients enrolled in the study.

Patient selection Patients ages 12-18 presenting to the emergency department with a mild traumatic brain injury and GCS >13 meeting inclusion criterial will be provided a study participation form to receive informed consent. ED staff will assess the patient's symptom severity with the Concussion Symptom Severity Score listed below. After this ED staff will assess the patient for inclusion criteria, followed by a healthcare provider Exclusion criteria will be evaluated by the healthcare provider at this time, and medical therapy can be initiated.

Inclusion criteria

* Age 12 to 18 years
* Presenting chief complaint of headache, head injury, or concussion following injury to the patient above the clavicles, within the first 48 hours of injury.
* GCS > 13 on arrival.

Exclusion criteria

* Age < 12 years or > 18 years
* Inability to provide informed consent
* Vomiting > 2 episodes following injury
* Physical or mental disability hindering adequate response to assessment of symptoms
* Hemodynamic instability/medical condition requiring further acute life-saving medical intervention
* Known brain mass, intracranial hemorrhage, skull fracture
* Known contraindications to magnesium use
* Known contraindication to Zofran use

Interventions Informed consent will be obtained after initial assessment of the patient by the healthcare provider, and inclusion/exclusion criteria are met.

After informed consent is obtained, and the patient meets the criteria for further acceptance into the study, then the patient's current symptoms will be screened by the healthcare providers. This will be the symptom score at time "0". After this the participants will receive 1 of 2 therapies that will be randomized by date of service whether it is an odd or even date. The treatment arm of the study (Even Days) will include 800mg of oral magnesium oxide along with a 4mg Zofran ODT as an initial dose in the emergency department. These participants will then continue to take 2 tablets of prescribed Magnesium oxide 400mg daily until their follow up with a physician at a local sports medicine clinic. The placebo arm (Odd days) of the study will receive 650 mg Acetaminophen, and a 4mg Zofran ODT in the emergency department. These participants continue to take scheduled acetaminophen 500 mg q8hr until follow up with a physician in the sports medicine clinic. The participants will have their symptom score re-evaluated after 1 hour of observation. If stable they will be discharged. A 24 hour follow up phone conversation will be placed by the primary investigators for a repeat of their symptom severity score. Finally, the participant will follow up in the outpatient sports medicine concussion clinic at 120 hours where a 4th symptom severity score will be obtained. These data will be collected and analyzed to compare the overall change in symptom severity score between the two treatment arms. The Aim of this study is to have a total n > 76. This will likely require 2 years of data collection. Our primary endpoint will be to evaluate if magnesium has an impact on participant's post-concussion severity index and a change in symptom severity score over time.

Symptom assessment Symptom assessment primarily described above, the investigators will use the standardized Post Concussion Severity. If the participant continues to have pain and a further intervention is required outside of the treatment and placebo arm the investigators will provide Ibuprofen weight adjusted for the participant's weight.

ED staff will re-assess the participant and record level of pain at time of study drug administration and at 60 minutes after study drug administration.

Data collection Primary data collection through the Concussion symptom severity index. Outcome measures Primary outcome is a comparison between the treatment and placebo groups in their changes in symptom severity scores over a 5-day period. Secondary endpoints include development of adverse effects related to medication administration, need for further intervention in the emergency department, and whether the participant's have returned to their baseline function by 120 hours.

Data analysis To be coordinated with Dr. William Corser, and an associated statistician team through Michigan State University. The study design will be a randomized cohort, repeat-measures efficacy study. The analysis of study results will look at data categorically, involving case or control group, and will also evaluate symptom scores at set intervals. An independent sample t test comparing the mean symptom severity scores among the cases and control groups at initial time of entry into the study, followed by repeat measurements after 1 hour, 24 hours and 120 hours will then be conducted. Point biserial correlation testing will also be employed to measure the strength of the relationship between being a member of either the case or control group with symptom severity scores. The primary outcome of this study will be the comparison of symptom severity scores between the treatment and placebo groups over a 5-day period. Anticipated secondary outcomes include but are not limited to adverse effects relating to medications administered, need for further intervention in the emergency department and return to baseline function within 120 hours.

Ethical Considerations Risks The risks of this study are minimal and related to the administration of medications. Acetaminophen, Zofran, and magnesium have low risk for development of adverse effects.

If an adverse reaction to these medications is to occur, while unlikely, the participant will be treated for these reactions symptomatically. Further medication administration will be based on the ED provider's discretion at the current standard of care and the participant's reactions will be documented/included in the secondary outcomes of the study.

Benefits Participant benefits include potential decreased duration of symptoms in the acute phase of injury following concussion. Magnesium is a relatively benign medication that is used frequently, and if this can contribute positively to acute concussion management, the investigators hope to change how mild traumatic brain injuries are managed.

Risk/benefit ratio Benefits of subject participation outweighs risk. Current standard of care is symptomatic care with rest, and follow up if symptoms persist 5-7 days following initial intervention. Adding magnesium, which has a low adverse effect profile and is an inexpensive option that could have a large impact on concussion management.

Participation Duration Participation in the proposed study will last the duration of their emergency department visit. Participation will involve a minimum of 30-60 minutes. The continued participation through the next 5 days is critical to the study to allow proper follow up, along with medication dosing.

Rationale for the use of selected subject population Concussions are a growing problem with socialization and media attention nationally. While there are no long term effects of concussions, there is an acute phase of injury that if decreased would benefit those with mild traumatic brain injury. With adolescents, there is a drive to return to normal health, and often an immediacy for treatment allowing appropriate initial intervention and follow up in the outpatient office prior to returning to daily activities. The interventions proposed in this study contain the current standard of care, thereby the addition of magnesium supplementation is medically benign but could have physiologic potential.

ELIGIBILITY:
Inclusion Criteria:

* • Age 12 to 18 years
* • Presenting chief complaint of headache, head injury, or concussion within the first 48 hours of injury.
* • GCS > 13 on arrival.

Exclusion Criteria:

* • Age < 12 years or > 18 years
* • Inability to provide informed consent
* • Vomiting > 2 episodes following injury
* • Physical or mental disability hindering adequate response to assessment of symptoms
* • Hemodynamic instability/medical condition requiring further acute life-saving medical intervention
* • Known brain mass, intracranial hemorrhage, skull fracture
* • Known contraindications to magnesium use
* • Known contraindication to Zofran use

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Change in symptom severity score | 4 scores total, time 0, time 1 hour, time 24 hours, time 120 hours
  Using post concussion symptom severity scores, the patient will complete symptom severity scores at specified intervals for comparison in post concussion severity score reduction. Higher scores indicate more severe symptoms, and lower scores indicate less severe symptoms.Post-Concussion Symptom Checklist Rating Mild Mod. Severe Initial 1 Hr. 48 Hr. 120 Hr. Headache 0-6 Nausea 0-6 Vomiting 0-6 Balance Problems 0-6 Dizziness 0-6 Visual Problems 0-6 Fatigue 0-6 Sensitivity to light 0-6 Sensitivity to noise 0-6 Numbness or Tingling 0-6 Pain other than Headache 0-6 Feeling as if "in a fog" 0-6 Feeling Slowed Down 0-6 Difficulty concentrating 0-6 Difficulty remembering 0-6 Drowsiness 0-6 Sleeping less than usual 0-6 Sleeping more than usual 0 1 2 3 4 5 6 Trouble falling asleep 0 1 2 3 4 5 6 More emotional than usual 0-6 Irritability 0-6 Sadness 0-6 Nervousness 0-6 Total Score

SECONDARY OUTCOMES:
Adverse events in the emergency department | 5 days
  Patients who require further treatment in the ED, require further medications, or develop adverse effects to the medications prescribed.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Trigger, MD, CAQSM, Principal Investigator — Lakeland Regional Health System
Locations (1):
- Lakeland Regional Healthcare, Saint Joseph, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller JW, D'Ambrosio R. When basic research doesn't translate to the bedside--lessons from the magnesium brain trauma study. Epilepsy Curr. 2007 Sep-Oct;7(5):133-5. doi: 10.1111/j.1535-7511.2007.00201.x. No abstract available. PMID 17998974
- [Background] Arango MF, Bainbridge D. Magnesium for acute traumatic brain injury. Cochrane Database Syst Rev. 2008 Oct 8;(4):CD005400. doi: 10.1002/14651858.CD005400.pub3. PMID 18843689
- [Background] Sen AP, Gulati A. Use of magnesium in traumatic brain injury. Neurotherapeutics. 2010 Jan;7(1):91-9. doi: 10.1016/j.nurt.2009.10.014. PMID 20129501
- [Background] Heath DL, Vink R. Concentration of brain free magnesium following severe brain injury correlates with neurologic motor outcome. J Clin Neurosci. 1999 Nov;6(6):505-9. doi: 10.1016/s0967-5868(99)90011-5. PMID 18639191
- [Background] Temkin NR, Anderson GD, Winn HR, Ellenbogen RG, Britz GW, Schuster J, Lucas T, Newell DW, Mansfield PN, Machamer JE, Barber J, Dikmen SS. Magnesium sulfate for neuroprotection after traumatic brain injury: a randomised controlled trial. Lancet Neurol. 2007 Jan;6(1):29-38. doi: 10.1016/S1474-4422(06)70630-5. PMID 17166799
- [Background] Zhao L, Wang W, Zhong J, Li Y, Cheng Y, Su Z, Zheng W, Guan XD. The effects of magnesium sulfate therapy after severe diffuse axonal injury. Ther Clin Risk Manag. 2016 Sep 27;12:1481-1486. doi: 10.2147/TCRM.S109482. eCollection 2016. PMID 27729796
- [Background] Heath DL, Vink R. Traumatic brain axonal injury produces sustained decline in intracellular free magnesium concentration. Brain Res. 1996 Oct 28;738(1):150-3. doi: 10.1016/0006-8993(96)00957-2. PMID 8949939
- [Background] Giza CC, Hovda DA. The new neurometabolic cascade of concussion. Neurosurgery. 2014 Oct;75 Suppl 4(0 4):S24-33. doi: 10.1227/NEU.0000000000000505. PMID 25232881
- [Background] McIntosh TK, Faden AI, Yamakami I, Vink R. Magnesium deficiency exacerbates and pretreatment improves outcome following traumatic brain injury in rats: 31P magnetic resonance spectroscopy and behavioral studies. J Neurotrauma. 1988;5(1):17-31. doi: 10.1089/neu.1988.5.17. PMID 3193462
- [Background] Hoane MR. Assessment of cognitive function following magnesium therapy in the traumatically injured brain. Magnes Res. 2007 Dec;20(4):229-36. PMID 18271492
- [Background] Busingye DS, Turner RJ, Vink R. Combined Magnesium/Polyethylene Glycol Facilitates the Neuroprotective Effects of Magnesium in Traumatic Brain Injury at a Reduced Magnesium Dose. CNS Neurosci Ther. 2016 Oct;22(10):854-9. doi: 10.1111/cns.12591. Epub 2016 Jul 15. PMID 27421816
- [Background] Cernak I, Vink R, Zapple DN, Cruz MI, Ahmed F, Chang T, Fricke ST, Faden AI. The pathobiology of moderate diffuse traumatic brain injury as identified using a new experimental model of injury in rats. Neurobiol Dis. 2004 Oct;17(1):29-43. doi: 10.1016/j.nbd.2004.05.011. PMID 15350963
- [Background] McKee JA, Brewer RP, Macy GE, Borel CO, Reynolds JD, Warner DS. Magnesium neuroprotection is limited in humans with acute brain injury. Neurocrit Care. 2005;2(3):342-51. doi: 10.1385/NCC:2:3:342. PMID 16159086
- [Background] Vollmer BL, Kirkwood MW, Comstock RD, Currie D, Grubenhoff JA. Assessing the Clinical Utility of the Question, "Is Your Child/Are You Back to Normal?" in Pediatric Concussion Symptom Resolution. Clin Pediatr (Phila). 2018 Feb;57(2):146-151. doi: 10.1177/0009922817693300. Epub 2017 Feb 15. PMID 28198194
- [Background] Randolph C, Millis S, Barr WB, McCrea M, Guskiewicz KM, Hammeke TA, Kelly JP. Concussion symptom inventory: an empirically derived scale for monitoring resolution of symptoms following sport-related concussion. Arch Clin Neuropsychol. 2009 May;24(3):219-29. doi: 10.1093/arclin/acp025. Epub 2009 Jun 23. PMID 19549721
- [Result] Li W, Bai YA, Li YJ, Liu KG, Wang MD, Xu GZ, Shang HL, Li YF. Magnesium sulfate for acute traumatic brain injury. J Craniofac Surg. 2015 Mar;26(2):393-8. doi: 10.1097/SCS.0000000000001339. PMID 25723660
- See also: Zofran FDA label — http://www.accessdata.fda.gov/drugsatfda_docs/label/2011/020103s030,020605s014,020781s014lbl.pdf